CLINICAL TRIAL: NCT04298281
Title: Testing Criteria for Convening Family Care Conferences in the Pediatric Intensive Care Unit
Brief Title: Family Care Conferences Criteria in the Pediatric Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: Advocate Lutheran General Hospital (Other); Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Kelly Michelson, Attending Physician, Ann & Robert H. Lurie Children's Hospital of Chicago, Ann & Robert H Lurie Children's Hospital of Chicago
Other Study IDs: 2020-3240
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Critical Illness
Keywords: Pediatrics; Family Care Conferences; Family Meetings
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents of patients who have a family care conference criteria: These will be parents of patient who have one of our defined family care conference criteria
- Parents of patients who do not have a family care conference criteria: These will be parents of patients who do not have one our defined family care conference criteria

SUMMARY:
Multidisciplinary experts from two Pediatric Intensive Care Units (PICUs), used an iterative modified Delphi process to develop and refine criteria for determining PICU patients for whom a family care conference would be beneficial. In this study the investigators will assess the use of those criteria as a trigger to offer parents of PICU patients a family care conference.

DETAILED DESCRIPTION:
Multidisciplinary experts from two Pediatric Intensive Care Units (PICUs) used an iterative modified Delphi process to develop and refine criteria for determining PICU patients for whom a family care conference would be beneficial. A preliminary set of criteria were developed with expert input and review of the literature. The investigators then assessed the preliminary criteria by retrospectively reviewing PICU patient's medical records at the two participating sites. Making revisions as needed the investigators then assessed the reliability of the family care conference criteria by prospectively reviewing the medical records of two months of PICU patient admissions at both participating sites. Based on these efforts, the investigators have described a set of family care conference criteria that will be studied in this investigation.

Primary Aim: Assess the inclusivity of the developed Family care conference criteria (FCC).

Secondary Aim: Describe parents' views of PICU family care conferences (FCC) and factors associated with having PICU family care conferences.

Methods: Taking an implementation science approach, the investigators will use plan-do-study-act cycles to optimize the goal of offering an FCC to all parent(s) of patients with any FCC criteria. The implementation aim statement is, within 6 months, healthcare team members will offer an FCC to the parent(s) of >95% of patients who have at least one FCC criteria.

* Planning (Plan). Development teams at participating institutions have determined how to inform PICU healthcare team members (HTMs) when a patient has an FCC criterion. A one-page information sheet (written at a 6th-grade level) describing FCCs, their potential role and value will be used when offering families a FCC. The development teams have also created an electronic health record (EHR) note template to document offering and conducting FCCs.
* Implementation (Do). Each weekday, a study team member at each site will review the EHR to identify patients who have one FCC criteria. A study team member will inform the PICU team when a patient has at least one FCC criteria and request that an HTM give the parent(s) the FCC information sheet, offer the parent(s) an FCC, and document the conversation with the parent(s) in the EHR. The processes for organizing and conducting FCCs will occur according to the PICU teams' discretion.
* Data collection (Study). The investigators will track the occurrence of FCCs by reviewing the EHR and obtaining input from PICU HTMs. For patients meeting at least one FCC criteria, but for whom an FCC was not documented, a study team member will ask the patient's PICU team (either resident, fellow, APRN, or attending) if an FCC occurred while the patient was admitted. For patients meeting FCC criteria, but for whom an FCC did not occur, study team members will also document if an FCC was offered by reviewing the EHR. If there is no EHR documentation about offering parent(s) an FCC, a study team member will ask the patient's PICU team (within a week of informing them that a patient met an FCC criteria) if the parent(s) were offered an FCC and if not why the parent(s) were not offered and FCC. Using input from HTMs, the investigators will record reasons for not offering an FCC and ascertain why parents opted out of an FCC. In addition to data about the FCC criteria, the investigators will extract the follow patient data from the EHR: age; sex; Pediatric Index of Mortality 3 (PIM3) score (measures of PICU admission illness severity) indication for PICU admission; need for intubation; need for pressors/vasoactive medications; number of subspecialty teams consulted; and use of ECMO.
* Revise implementation plan (Act). The development teams will meet every other week x 4, then monthly x 4, then every two months to review the data, assess implementation, and modify the process as needed.

To describe parents' views of PICU FCCs and factors associated with having PICU FCCs, the investigators will enroll English- and Spanish-speaking (materials will be available in Spanish) parents (one or both) of PICU patients <18 years old for whom an FCC occurred or whose child had at least one FCC criteria. English- and Spanish-speaking parents (one or both) of PICU patients < 18 years old whose child did not have an FCC criteria and who did not have an FCC will also be eligible until the investigators have enrolled 100 parents. the investigators will invite eligible parents to complete a post-FCC Survey within three days of an FCC (for those that have an FCC). The investigators will invite all eligible parents to complete a post-PICU Survey and participate in a one-on-one interview within three days of PICU discharge.

The Post-FCC Survey will ask for information about parent characteristics and feedback on the FCC. The variables related to parent characteristics will include demographics, family relationship style (using the Family Apgar), informational support (using the Informational Support SF4a), and mental health (using the two-item PROMIS® mental health scale) and global physical health (using the two-item PROMIS® global physical health scale). Items asking for feedback about the FCC (adapted from previous work) will assess: overall FCC utility; the topics discussed and their importance to the parents; what was useful and what could be improved; and whether the parent would like to have another FCC in the future. The post-PICU Survey will include the same items asking about family characteristics as in the Post-FCC Survey (not included for parents who completed a post-FCC Survey). The post-PICU Survey will also include items asking about the utility of other modes of PICU communication (daily rounds, electronic patient portals, written information, bedside and phone interactions with physicians/APRNs and bedside nurses, and communication with social workers, chaplains, and case managers). Finally, the post-PICU Survey will ask if an FCC was offered, request feedback on FCCs (see above) that occurred (not included if a post-FCC Survey was completed), and ask why offered FCCs did not occur. All non-validated survey items were reviewed by the study team, for face validity. Parents of patients who die in the PICU will receive the post-PICU Survey by mail or email 3-5 weeks after their child's death, as the investigators and others have done previously. Parents will complete surveys electronically on a tablet using REDCap. Audio-recorded one-on-one interviews will be conducted by a study team member using an interview guide that focuses on the following content areas: perceptions of PICU communications overall; specific modes of communication; why an FCC occurred or did not occur; and perceptions of FCC utility.

ELIGIBILITY:
Inclusions criteria:

* All parents of patients < 18 years old in the PICU during the study time period.
* Parents who are English or Spanish speakers
* Parents who agree to participate by completing the questionnaire
* Parents who agree to participate in the recorded interview by completing the interview

Exclusion criteria:

• None

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: * Pediatric Intensive Care Unit Patients
  * Parents of Pediatric Intensive Care Unit Patients
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Family Care Conference Criteria Sensitivity | Through PICU admission, an average of 3.5 days and up to 3 months
  Sensitivity of our Family Care Conference Criteria. Sensitivity can range from 0% - 100%

SECONDARY OUTCOMES:
Parents' views of PICU Family care conference based on survey responses | Through PICU admission, an average of 3.5 days and up to 3 months
  We will describe parents' views of PICU Family Care conferences based on responses to a survey developed with expert input and existing literature.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly N Michelson, MD, MPH, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (2):
- United States (2):
  - Ann Robert Lurie children's hospital, Chicago, Illinois
  - Advocate Lutheran General Children's Hospital, Park Ridge, Illinois

IPD SHARING:
Plan to Share IPD: Undecided
undecided at this moment